CLINICAL TRIAL: NCT00158509
Title: Efficacy of an HSV2 Genital Herpes Suppressive Treatment on HIV and HSV2 Genital Shedding Among Co-Infected Patients Receiving or Not Antiretroviral Drugs
Brief Title: Randomised Controlled Trial Assessing the Impact of Genital Herpes Suppressive Therapy on HIV Shedding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANRS 1285
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-06-07 (Estimated); Status verified 2006-06

CONDITIONS: Herpes Genitalis; HIV Infection
Keywords: Valacyclovir; HIV-1; HSV-2; genital shedding; herpes genitalis; HIV infection
MeSH Terms: conditions — Herpes Genitalis; HIV Infections | interventions — Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir

SUMMARY:
Genital herpes is a long-life sexually transmitted diseases which infects a large proportion of women in Africa. Its clinical symptoms are painful sores on the genitals, which heals after a few days. HIV infection can worsen genital herpes. In turn, it is possible that genital herpes increases the quantity of HIV secreted at the genital level in women infected by the 2 viruses. This study is dedicated to verify this hypothesis.

DETAILED DESCRIPTION:
Infection with Herpes Virus Simplex type 2 (HSV-2) is likely to represent the main cofactor involved in HIV transmission, either through clinical episodes or asymptomatic genital shedding. However, the definite proof of this concept has never been made through randomised controlled trials. Furthermore, the natural history of HSV-2 infection is poorly documented in sub-Saharan Africa, as well as the efficacy of the antiviral drug on virus transmission. The latter can be measured by HSV-2 genital shedding as a proxy.

The objectives of this research programme are to assess the impact of a suppressive treatment for genital herpes on HIV genital shedding among co-infected patients receiving HAART or not needing antiretroviral (ARV) drugs.

In order to achieve these objectives, we propose to perform 2 randomised double blind controlled trials nested within the ongoing cohort of sex workers in Bobo-Dioulasso.

While the increase of HIV transmission by HSV-2 infection stands as our main working hypothesis among HIV positive persons, the specific rationale for individuals taking ARV is the following: Does the potential cofactor effect of genital herpes on HIV remain present when the immunity is built up by ARV? In other words, is HSV-2 infection a public health issue in this group of people. The role of ARV on HIV transmission will also be assessed.

These 2 trials will be performed using exactly the same methodology and the same study treatment. We will use a parallel design with a baseline phase to take into account the important inter-individual variability of genital shedding. Each participant will be its own control. The baseline phase and treatment phases will each consist of 6 visits performed at a 2 weeks interval. The participants will receive either placebo or Valacyclovir 1g/day during the treatment phase (3 months).

The outcomes will be measured using both a qualitative and a quantitative measure of HIV shedding. The analysis will be conducted using an "intention to treat" and a "per protocol" approach.

At the end of our project, the working hypothesis will be much documented in women taking ARV or not. Furthermore, our results will constitute a reference for an upcoming therapeutic vaccine trial.

This work results from the collaboration of the Centre Muraz, the UMR 36 "AIDS and associated diseases" (Montpellier) and the London School of Hygiene & Tropical Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Infection with HIV-1 and HSV-2
* If required to take antiretrovirals according to WHO recommendations, should be on HAART for at least 4 months
* Written informed consent

Exclusion Criteria:

* Pregnancy or willing to be pregnant during the next 6 months
* Breastfeeding
* Renal failure
* Expected non-compliance with follow-up or study treatment

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215
Dates: Start 2004-08; Study Completion 2005-07

PRIMARY OUTCOMES:
To assess the impact of HSV-2 suppressive therapy on HIV shedding among co-infected women taking highly active antiretroviral therapy (HAART) or not needing HAART

SECONDARY OUTCOMES:
To assess the impact of HSV-2 suppressive therapy on HSV-2 shedding among co-infected women taking HAART or not needing HAART

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Nagot, Principal Investigator — London School of Hygiene and Tropical Medicine; Philippe Mayaud, Study Chair — London School of Hygiene and Tropical Medicine; Philippe Van de Perre, Study Chair — Montpellier University, France
Locations (1):
- Service d'Hygiene du Centre Muraz, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Result] Nagot N, Foulongne V, Becquart P, Mayaud P, Konate I, Ouedraogo A, Defer MC, Weiss H, Van de Perre P, Segondy M. Longitudinal assessment of HIV-1 and HSV-2 shedding in the genital tract of West African women. J Acquir Immune Defic Syndr. 2005 Aug 15;39(5):632-4. PMID 16044019
- [Derived] Mayaud P, Nagot N, Konate I, Ouedraogo A, Weiss HA, Foulongne V, Defer MC, Sawadogo A, Segondy M, Van de Perre P; ANRS 1285 Study Group. Effect of HIV-1 and antiretroviral therapy on herpes simplex virus type 2: a prospective study in African women. Sex Transm Infect. 2008 Oct;84(5):332-7. doi: 10.1136/sti.2008.030692. Epub 2008 Jul 2. PMID 18596069
- [Derived] Nagot N, Ouedraogo A, Konate I, Weiss HA, Foulongne V, Defer MC, Sanon A, Becquart P, Segondy M, Sawadogo A, Van de Perre P, Mayaud P; ANRS 1285 Study Group. Roles of clinical and subclinical reactivated herpes simplex virus type 2 infection and human immunodeficiency virus type 1 (HIV-1)-induced immunosuppression on genital and plasma HIV-1 levels. J Infect Dis. 2008 Jul 15;198(2):241-9. doi: 10.1086/589621. PMID 18593294
- [Derived] Nagot N, Ouedraogo A, Foulongne V, Konate I, Weiss HA, Vergne L, Defer MC, Djagbare D, Sanon A, Andonaba JB, Becquart P, Segondy M, Vallo R, Sawadogo A, Van de Perre P, Mayaud P; ANRS 1285 Study Group. Reduction of HIV-1 RNA levels with therapy to suppress herpes simplex virus. N Engl J Med. 2007 Feb 22;356(8):790-9. doi: 10.1056/NEJMoa062607. PMID 17314338